CLINICAL TRIAL: NCT04320940
Title: A Randomized, Double-Blind, Controlled Study to Assess the Efficacy and Safety of Intravenous Phenobarbital in Neonatal Seizures
Brief Title: Efficacy and Safety of Intravenous Phenobarbital in Neonatal Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient participant recruitment hindered the study's progress, preventing robust data collection and compromising statistical power
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MI-5780
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy, Benign Neonatal
Keywords: Neonatal Seizures; Phenobarbital; Anticonvulsants
MeSH Terms: conditions — Epilepsy, Benign Neonatal | interventions — Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phenobarbital Sodium Injection 20mg (Active Comparator): Following confirmation of seizure criteria and randomization, subjects will receive Phenobarbital 20 mg/kg (first/initial dose) followed by 20 mg/kg (if required).
  Interventions: Drug: Phenobarbital Sodium Injection
- Phenobarbital Sodium Injection 40mg (Active Comparator): Following confirmation of seizure criteria and randomization, subjects will receive Phenobarbital 40 mg/kg (first/initial dose) followed by 10 mg/kg (if required).
  Interventions: Drug: Phenobarbital Sodium Injection

INTERVENTIONS:
Drug: Phenobarbital Sodium Injection — The initial dose will be administered intravenously over a 30-minute period. The time period between the first and second dose of phenobarbital cannot occur within 30 minutes of the end of the first dose.
  Other Names: Phenobarbital

SUMMARY:
This is a randomized, double-blind, parallel-group, Phase 3 study to evaluate the efficacy of the administration of phenobarbital sodium injection in neonates who have suffered from electrographic or electroclinical seizure. As neonatal seizures can have long-term adverse effects, including death, placebo-controlled studies are not appropriate for this population. This study is designed to show intravenous phenobarbital is effective at preventing subsequent seizures by demonstrating greater efficacy at a higher dose compared to a lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female neonates with a gestational age of ≥ 34 - ≤44 weeks admitted into the NICU with a high probability of developing seizures (e.g., HIE, stroke, intracerebral hemorrhage, central nervous system infection)
* Parental informed consent (in-person or remote consent)
* Undergoing continuous video electroencephalogram (cvEEG) monitoring
* Has evidence of electrographic seizure burden of at least 30 seconds/h

Exclusion Criteria:

* Received anticonvulsant treatment, including phenobarbital, prior to randomization (with exception of lorazepam administered for sedation > 24 hours before enrollment)
* Strong suspicion or confirmed diagnosis of brain malformation, inborn error of metabolism genetic syndrome, or major congenial malformation prior to randomization
* Seizures responding to correction of hypoglycemia, hypocalcemia or any other metabolic disorder
* Death appears to be imminent as assessed by the NICU attending physician
* Is currently enrolled in another study assessing the same and/or similar primary/secondary endpoints with/without drug treatment.

Ages: 34 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pergolizzi Jr., MD, MD, Principal Investigator — NEMA Research, Inc.
Locations (8):
- United States (7):
  - Arkansas Cildren's Hospital, Little Rock, Arkansas
  - Children's National Hospital, Washington D.C., District of Columbia
  - South Miami Hospital, Miami, Florida
  - Jamie Flores-Torres, Tampa, Florida
  - Matthew Butoryak, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Marshall Health, Huntington, West Virginia
- Jordan University of Science and Technology (King Abdullah University Hospital, KAUH), Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Neonates Who do Not Require Additional Seizure Treatment After the First Dose of Phenobarbital.
Description: Percent of neonates who do not require additional seizure treatment after the first dose of phenobarbital during the first 24 hours after treatment.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
Number analyzed (Participants) | 3 | 1
Participants | 2 | 1

2. Secondary Outcome: Neonates Who do Not Require Additional Seizure Treatment After the First Dose of Phenobarbital.
Description: Percent of neonates who do not require additional seizure treatment after 2 hours of the first dose of phenobarbital.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
Number analyzed (Participants) | 3 | 1
Participants | 2 | 1

3. Secondary Outcome: Neonates Who do Not Require Additional Seizure Treatment After the Second Dose of Phenobarbital.
Description: Percent of neonates who do not require additional seizure treatment after the second dose of phenobarbital within the first 24 hours of treatment.
Time Frame: 24 hours
Population: Three subjects (two in the low-dose and one in the high-dose groups) received a first dose and no subsequent doses of the medication. One subject in the low-dose group received an initial dose (20 mg/kg) at 14:10 on July 15 and a second dose (20 mg/kg) at 17:25 on the same day.
Measure: Count of Participants; unit: Participants
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

4. Secondary Outcome: Seizure Burden Over 48 Hours Following Initial Administration of the Phenobarbital Injection.
Description: Number of subject required monitoring of seizure burden over 48 hours following initial administration of the phenobarbital injection.
Time Frame: 48 hours
Population: One subject in the low-dose group received an initial dose (20 mg/kg) at 14:10 on July 15 and a second dose (20 mg/kg) at 17:25 on the same day. Maintenance doses of 5 mg/kg were administered to this subject once daily on July 16, 17, and 18. Only this subject required monitoring of seizure burden over 48 hours following initial administration of the phenobarbital injection
Measure: Count of Participants; unit: Participants
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Serious Adverse Events were assessed up to 30 days following the first treatment, on average 45 days. Other (Not Including Serious) Adverse Events were assessed for up to 24 hours following the first treatment and up to 4 days.
Arm/Group | Phenobarbital Sodium Injection 20mg | Phenobarbital Sodium Injection 40mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenobarbital Sodium Injection 20mg (N=3) | Phenobarbital Sodium Injection 40mg (N=1)
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — One subject (1 Group A) experienced one TEAE of moderate pulmonary hypertension. This TEAE was not expected, not related to the study drug, and resolved in 21 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04320940/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04320940/SAP_001.pdf